CLINICAL TRIAL: NCT00387894
Title: Phase-2 Study of Tarceva in Patients With Recurrent EGFR Positive and Phosphatase and Tensin Homolog (PTEN) Wild Type Glioblastoma Multiforme and Gliosarcoma
Brief Title: Erlotinib in Treating Patients With Recurrent Glioblastoma Multiforme or Gliosarcoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient accrual of population likely to benefit; progression in 6 patients
Sponsor: Michael Prados (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Michael Prados, Professor, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000492762; UCSF-06102 (Other: OnCore); UCSF-H5941-28905-01 (Other: IRB Approval #); GENENTECH-OSI3765s (Other: Sponsor protocol ID)
Record Dates: First submitted 2006-10-12; First posted 2006-10-13 (Estimated); Results first posted 2013-05-17 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-04

CONDITIONS: Adult Brain Tumors
Keywords: adult glioblastoma; adult gliosarcoma; recurrent adult brain tumor
MeSH Terms: conditions — Brain Neoplasms; Glioblastoma; Gliosarcoma | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- erlotinib hydrochloride (Tarceva) (Experimental): During the treatment period, patients who are not receiving EIAED (Group A) will receive single-agent Tarceva, 150 mg/day. Patients on EIAED (Group B) will receive single-agent Tarceva, 600 mg/day. Tablets should be taken at the same time each day with 200 mL of water at least 1 hour before or 2 hours after a meal. Patients who are unable to swallow tablets may dissolve the tablets in distilled water for administration. The dose of Tarceva will be escalated after 14 days to 200 mg/day (Group A) or 650 mg/day (Group B) assuming no intolerable grade 2 rash, any grade 3 rash, or grade 2 diarrhea despite loperamide.
  Interventions: Drug: erlotinib hydrochloride

INTERVENTIONS:
Drug: erlotinib hydrochloride — Tarceva will be self-administered in an open-label, unblinded manner to all patients enrolled in the study. During the treatment period, patients who are not receiving EIAED (Group A) will receive single-agent Tarceva, 150 mg/day. Patients on EIAED (Group B) will receive single-agent Tarceva, 600 mg/day. Tablets should be taken at the same time each day with 200 mL of water at least 1 hour before or 2 hours after a meal. Patients who are unable to swallow tablets may dissolve the tablets in distilled water for administration. The dose of Tarceva will be escalated after 14 days to 200 mg/day (Group A) or 650 mg/day (Group B) assuming no intolerable grade 2 rash, any grade 3 rash, or grade 2 diarrhea despite loperamide.
  Other Names: Tarceva

SUMMARY:
RATIONALE: Erlotinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase II trial is studying how well erlotinib works in treating patients with recurrent glioblastoma multiforme or gliosarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the objective response rate in patients with recurrent epidermal growth factor receptor (EGFR)-positive and PTEN wild-type glioblastoma multiforme or gliosarcoma treated with erlotinib hydrochloride.

Secondary

* Assess the response rate in patients who also EGFRVIII mutant and PTEN wild type glioblastoma multiforme or gliosarcoma.
* Determine the progression-free survival of patients treated with this drug.

OUTLINE: This is an open-label study. Patients are stratified according to concurrent use of enzyme-inducing antiepileptic drugs (EIAEDs) (yes vs no).

Patients receive oral erlotinib hydrochloride once daily on days 1-28. Treatment repeats every 4 weeks for up to 1 year in the absence of disease progression or unacceptable toxicity. Some patients may receive additional erlotinib hydrochloride after 1 year at their physician's discretion.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study.

ELIGIBILITY:
INclusion Criteria:

* Diagnosis of glioblastoma multiforme (GBM) or gliosarcoma (GS)

  * In first, second, or third relapse
  * History of low-grade glioma with transformation to GBM or GS allowed

    * Considered to be in first relapse at first documented diagnosis of GBM or GS
* Measurable or evaluable disease by contrast MRI
* Must have failed prior treatment that included external beam radiotherapy with or without chemotherapy
* Epidermal growth Factor Receptor-positive and PTEN wild-type by immunohistochemistry

PATIENT CHARACTERISTICS:

* Karnofsky performance status 60-100%
* WBC ≥ 3,000/mm³
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 10 g/dL (transfusion allowed)
* SGOT < 2 times upper limit of normal (ULN)
* Bilirubin < 2 times ULN
* Creatinine < 1.5 mg/dL OR creatinine clearance ≥ 60 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective hormonal or barrier method contraception before, during, and for at least 12 weeks after completion of study treatment
* No other cancer within the past 3 years except nonmelanoma skin cancer or carcinoma in situ of the cervix
* No active infection
* No other disease that would obscure toxicity or dangerously alter study drug metabolism

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 4 weeks since prior and no concurrent radiotherapy
* At least 4 weeks since prior and no concurrent cytotoxic chemotherapy agents (e.g., temozolomide) (6 weeks for nitrosoureas)
* At least 2 weeks since prior and no concurrent noncytotoxic chemotherapy agents
* At least 4 weeks since prior investigational agents
* No other concurrent investigational agents
* No prior erlotinib hydrochloride or other epidermal growth factor receptor tyrosine-kinase inhibitors
* At least 2 weeks since prior enzyme-inducing antiepileptic drugs (EIAEDs), if not used concurrently with study treatment

  * Concurrent continuous use of EIAEDs allowed provided the patient has received the drug for ≥ 2 weeks prior to study treatment
* No concurrent immunotherapy or anticancer hormonal therapy
* No other concurrent antineoplastic or antitumor agents

Exclusion Criteria:

Patients meeting any of the following criteria are ineligible for study entry:

* Patients with a history of any other cancer (except non-melanoma skin cancer or carcinoma in-situ of the cervix), unless in complete remission and off of all therapy for that disease for a minimum of 3 years are ineligible.
* Patients must not have active infection
* Patients must not be pregnant/breast feeding and must agree to practice adequate contraception. Women of childbearing potential must have a negative B-HCG pregnancy test documented within 14 days prior to treatment. Patients must not be pregnant because of the uncertainty that study drug may be potentially embryotoxic. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry, for the duration of study participation, and continue approximately 12 weeks after the study is completed. If condoms are used as a barrier contraceptive, a spermicidal agent should be added to ensure that pregnancy does not occur. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Prior treatment with Tarceva, or other EGFR tyrosine-kinase inhibitors will not be allowed.
* Patients must not have any disease that will obscure toxicity or dangerously alter drug metabolism.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2007-01; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael D. Prados, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Oral Erlotinib Hydrochloride (Tarceva) Daily on Days 1-28: Tarceva self-administered in an open-label, unblinded manner to all patients enrolled. During the treatment period, patients who are not receiving enzyme-inducing antiepileptic drugs (EIAED) will receive single-agent Tarceva, 150 mg/day. Patients on EIAED will receive single-agent Tarceva, 600 mg/day. Tablets should be taken at the same time each day with 200 mL of water at least 1 hour before or 2 hours after a meal. Patients who are unable to swallow tablets may dissolve the tablets in distilled water for administration. The dose of Tarceva will be escalated after 14 days from 150 to 200 mg/day or from 600 to 650 mg/day assuming no intolerable grade 2 rash, any grade 3 rash, or grade 2 diarrhea despite loperamide.
Period: Overall Study
Arm/Group | Oral Erlotinib Hydrochloride (Tarceva) Daily on Days 1-28
Started | 6
Completed | 5
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Oral Erlotinib Hydrochloride (Tarceva) Daily on Days 1-28: erlotinib hydrochloride (Tarceva) self-administered in an open-label, unblinded manner to all patients enrolled in the study.
Arm/Group | Oral Erlotinib Hydrochloride (Tarceva) Daily on Days 1-28
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Age Continuous [Mean (Full Range); unit: years] | 44 [27 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Disease Response Measured Objectively by MRI of Brain
Description: Lack of disease progression indicates response to treatment
Time Frame: Every 8 weeks or as indicated
Population: 5 participants evaluable while receiving study treatment
Measure: Number; unit: participants
Arm/Group | Oral Erlotinib Hydrochloride (Tarceva) Daily on Days 1-28
Number analyzed (Participants) | 5
participants
  Disease progression prior to 8 weeks | 4
  Disease responsive at 8 Weeks | 1
  Disease responsive at 16 Weeks | 0

2. Secondary Outcome: Duration of Progress-free Survival (PFS)
Description: Patients with stable or responding disease will continue treatment until tumor progression is determined
Time Frame: Until first observation of progressive disease, non-reversible neurologic progression or permanently increased steroid requirement (stable disease only), death due to any cause (up to 16 weeks)
Measure: Number; unit: participants
Arm/Group | Oral Erlotinib Hydrochloride (Tarceva) Daily on Days 1-28
Number analyzed (Participants) | 5
participants
  2 weeks PFS | 1
  3 weeks PFS | 1
  6 weeks PFS | 2
  12 weeks PFS | 1

ADVERSE EVENTS:
Time Frame: 30 days after the last study treatment, thereafter for survival
Description: Only AEs Grade 3 or higher were required to be collected as AEs, per protocol
Arm/Group | Oral Erlotinib Hydrochloride (Tarceva) Daily on Days 1-28
Serious Adverse Events (participants affected / at risk) | 6/6
Other Adverse Events (participants affected / at risk) | 0/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Erlotinib Hydrochloride (Tarceva) Daily on Days 1-28 (N=6)
Disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) — All participants died due to disease progression
Neuropathy (Nervous system disorders) | 1 (1) — Grade 3, not related to treatment
Wound complication (Skin and subcutaneous tissue disorders) | 1 (1) — Grade 3, not related to treatment
Seizure (General disorders) | 1 (1) — Grade 3, not related to treatment
Confusion (General disorders) | 1 (1) — Grade 3, not related to treatment

LIMITATIONS AND CAVEATS:
The study was terminated early for 2 reasons: 1. ongoing literature at the time confirming that the selection process was not likely to enrich for a patient population expected to benefit, and 2. Rapid disease progression in the first 6 patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No